CLINICAL TRIAL: NCT03020290
Title: Long Superficial Femoral Artery Stenting With SuperA Interwoven Nitinol Stents
Acronym: STELLASUPERA
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: RC15_0464
Record Dates: First submitted 2016-12-21; First posted 2017-01-13 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2019-09

CONDITIONS: Atherosclerosis Obliterans
Keywords: femoropopliteal artery; interwoven nitinol stent; self-expanding-endovascular; TASC C and TASC D; Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with femoropopliteal lesion: patients with femoropopliteal lesion - Endovascular treatment for PAD during medical care
  Interventions: Device: Endovascular treatment for PAD during medical care (SuperA stent (Abbott))

INTERVENTIONS:
Device: Endovascular treatment for PAD during medical care (SuperA stent (Abbott)) — Long femoropopliteal stenting with SuperA devices during medical care. The endovascular treatment for PAD will be done during the usual medical treatment of patient. The intervention is not carried out within the framework of the research protocol
  Other Names: long femoropopliteal revascularization

SUMMARY:
Endovascular treatment with stenting is currently used in the treatment of femoro-popliteal lesions. This technique tends to extend to lesions for which the gold standard remains until now the open surgery treatment (lesions TASC C and D).

The primary objective of the study was to evaluate the clinical efficacy at 12 months of the SuperA stent (Abbott) in the treatment of long de novo atherosclerotic lesions TASC C and D in patients with symptomatic peripheral arterial disease. The secondary objectives are to evaluate the clinical effectiveness of the SuperA stent at 24 months, according to clinical, morphological and haemodynamic criteria, the possible influence of calcifications and the quality of life of patients.

The SuperA stent treatment is not specifically provided for by the Protocol but is carried out within the framework of the care. This study is an observationnal study.

DETAILED DESCRIPTION:
Patient will be recruiting during 1 year. Patient will be followed in the study during 2 years. Pre-operative exams are collected. Patients are asked to give their oral authorization to participate in the study by their surgeon.

Patient can be included up to the next day of the intervention.

Endovascular treatment of femoropopliteal lesion with SuperA stents during medical care:

Intervention will be achieved in operative room, under local anesthesia and sedation or general anesthesia. An angio-CT or an arteriography is necessary to attest the presence for TASC C or D lesion involving the superficial femoral and/or popliteal arteries.

The long femoropopliteal lesion must be pre-dilated during 3 minutes with a balloon of 1mm diameter more than the stent to be implanted.

A control arteriography will be done before the implantation of the stent and at the end of the intervention to assess the success of the procedure.

If needed, endovascular treatment could be realized on the inflow or outflow in the same time.

Patient follow-up :

Patient follow-up is performed at 1, 6, 12 and 24 months. Follow-up will systematically include a clinical evaluation and a duplex scan with the ankle brachial index (ABI).

The x-rays and the quality of life questionnaire will be done at 1, 12 and 24 months.

All clinical surveillance events, complications and re-hospitalizations will be collected.

ELIGIBILITY:
Inclusion criteria:

* Age > 18 years,
* Symptomatic PAD, Rutherford 2 to 6
* Atherosclerotic femoropopliteal lesion TASC C or D (on CT scan or arteriography)
* De novo femoropopliteal lesion
* Patient informed of the study and oral authorization collected

Exclusion Criteria:

* Under-age patient
* Patient of age, but under legal guardianship or care
* Potentially pregnant women
* Patients do not understand the French language
* Asymptomatic lesion
* Acute ischemia or acute thrombosis
* Lesion already treated
* No-atherosclerotic disease
* hemostasis disorder
* severe comorbidity with life expectancy less than 2 years
* contraindication of antiplatelet (dual antiplatelet therapy required during at least 2 month post-intervention)
* patient participating in a clinical trial likely to interfer
* Comorbidity or other, according investigator, that may interferer with the conduct of the study
* lesion near to an aneurysm
* Patient follow-up impossible
* Patient refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients included in this study are major patients and have lower limb arteriopathy requiring a therapeutic gesture in the femoro-popliteal segment. The inclusion in this study will be proposed to the patients during the consultation of preoperative vascular surgery or during the hospitalization, until the day after their intervention. The number of subjects planned is 50.
  In the case where the patient has bilateral femoropopliteal lesions, the limbs being treated in separate hospitalizations, both members may be treated with SuperA stents. The two members will then be considered independently of each other.
  Patients with associated lesions requiring treatment, any artery confused, may be treated at the same operative time if deemed necessary by the surgeon.
Sampling Method: Non-Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2016-12; Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
Number of patient with improvement of at least one category of Rutherford classification | 12 months
  To evaluate the sustained clinical effectiveness of the SuperA stent (Abbott) at 12-month for TASC C and D atherosclerotic femoropopliteal lesions in patients with symptomatic primary artery disease (PAD) (RUTHERFORD 2 to 6).
  Improvement of at least 1 category of Rutherford classification for claudicants.
  Healing of a trophic disorder and disappearance of resting pain for patient with critical ischemia

SECONDARY OUTCOMES:
Number of patient with improvement of at least one category of Rutherford classification | 24 months
  clinical effectiveness of the SuperA stent measurement
number of patient presenting a major adverse cardiovascular event | 24 months
  clinical effectiveness of the SuperA stent measurement
number of patient presenting a major adverse limb event | 24 months
  clinical effectiveness of the SuperA stent measurement
limb salvage rate measurement | 24 months
  clinical effectiveness of the SuperA stent measurement
rate of Target Lesion Revascularization (TLR) | 24 months
  Effectiveness of the SuperA stent measurement
rate of Target Extremity Revascularization (TER) | 24 months
  Effectiveness of the SuperA stent measurement
number of patient with sustained permeability without restenosis > 30% in lack of reintervention | 24 months
  hemodynamic effectiveness of the SuperA stent measurement
number of patient with sustained permeability without restenosis > 30% after reintervention | 24 months
  hemodynamic effectiveness of the SuperA stent measurement
variation of the ABI (Ankle systolic pression (mmHg) / brachial systolique pression (mmHg) index) before and after surgery | 24 months
  hemodynamic effectiveness of the SuperA stent measurement
  (restenosis, thrombosis) and morphologic criteria (stenting length, stent fracture).
restenosis measurement | 24 months
  hemodynamic effectiveness of the SuperA stent measurement
thrombosis measurement | 24 months
  hemodynamic effectiveness of the SuperA stent measurement
stenting length measurement | 24 months
  morphologic criteria of effectiveness of the SuperA stent measurement
stent fracture measurement | 24 months
  morphologic criteria of effectiveness of the SuperA stent measurement
quality of life in patients treated with the SuperA stent | 1 month
  EuroQol five dimensions questionnaire (EQ5D-3L)
quality of life in patients treated with the SuperA stent | 12 months
  EQ5D-3L questionnaire
quality of life in patients treated with the SuperA stent | 24months
  EQ5D-3L questionnaire
Assessment of vessel calcification rate | 24months
  For predictive factors of failure
Assessment of elongation rate of SuperA | 24months
  For predictive factors of failure
Assessment of stent diameter | 24months
  For predictive factors of failure
Number of patient presenting cardiovascular comorbidity | 24months
  For predictive factors of failure
Number of patient presenting a renal dysfunction (creatinine clearance < 60 mL/min and/or dialysis) | 24months
  For predictive factors of failure
Number of patient treated with anti-platelet therapy | 24months
  For predictive factors of failure

CONTACTS AND LOCATIONS:
Overall Officials: Yann Goueffic, PU-PH, Principal Investigator — yann.goueffic@chu-nantes.fr
Locations (2):
- France (2):
  - CHD Vendée, La Roche-sur-Yon
  - Nantes CHU, Nantes